CLINICAL TRIAL: NCT01051830
Title: A Care Model for Hip-fractured Elderly Persons With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Yea-Ing Lotus Shyu, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NHRI-EX103-9905PI; CGMH-98-0327B (Other: Chang Gung Memory Hospital, Taiwan)
Record Dates: First submitted 2010-01-17; First posted 2010-01-20 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes Mellitus; Hip Fracture
MeSH Terms: conditions — Diabetes Mellitus; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interdisciplinary group (Experimental): Diabetes intervention and rehabilitation program. The rehabilitation program includes geriatric consultation, the rehabilitation program (interventions to improve ROM, muscle strength and endurance, proprioceptive enhancement, balance capacity, aerobic and anaerobic capacity, flexibility, and body composition), and discharge-planning services. The DM intervention includes: dietary and DM education, blood pressure control, dyslipidemia management, a glycemic treatment regimen, and exercises.
  Interventions: Other: Diabetes interdisciplinary program
- Control group (No Intervention): Routine care

INTERVENTIONS:
Other: Diabetes interdisciplinary program — Diabetes consulting, rehabilitation program
  Arms: Interdisciplinary group

SUMMARY:
The purpose of this study is to 1) develop a well-conceived and feasible protocol for hospital discharge and subacute care for hip-fractured elderly persons with DM, and 2) compare the costs and effectiveness of this DM-specific model with those of an effective subacute care model previously developed by our research team.

DETAILED DESCRIPTION:
Clinical and scientific significance. Health outcomes, as well as physical and cognitive function, have been shown to be negatively impacted by comorbidity beyond the bare sum of effects due to the single diseases. One such comorbidity is diabetes mellitus (DM), a global health issue and the fifth major cause of death in Taiwan from 1987 to 2001. Starting in 2002, DM has become the fourth. Hip-fractured elderly persons with DM were shown in our previous studies to have significantly higher mortality and readmission rates and poorer recovery in walking ability and various physical health outcomes than those without DM during the first year after discharge. Clinical evidence has shown that elderly patients with hip fracture can benefit from postoperative rehabilitation, early discharge-planning programs, or transitional care programs. However, little is known about effective interventions specifically for hip fractured patients with DM.

Research Purposes. The purpose of this study is to 1) develop a well-conceived and feasible protocol for hospital discharge and subacute care for hip-fractured elderly persons with DM, and 2) compare the costs and effectiveness of this DM-specific model with those of an effective subacute care model previously developed by our research team.

Data and Methods. A clinical trial with 1-year follow-up will be used to compare the cost-effectiveness of the DM-specific model in 88 hip-fractured elderly patients with that of our subacute care model (n=88) and routine care (n=88). Patients will be recruited through the emergency room of Chang Gung Memorial Hospital (CGMH) at Lin Kuo. Subjects will be assessed before surgery, before discharge, at 1, 3, 6, and 12 months after discharge for biometric measures, DM-related outcomes, clinical outcomes, self-care ability, health-related quality of life, service utilization, and costs of care. To maximize outcomes sensitive to the intervention, biometric measures of activity will be included, i.e., daily energy consumption and arterial stiffness index. DM-related variables will include haemoglobin A1c (HbA1c), tendon reflexes, superficial and deep sensation, peripheral pulses, diabetic retinopathy, signs of "diabetic foot," use of medication, and clinical procedures. The study has already been approved by the Institutional Review Board of CGMH. Trajectories of the outcome variables and their predictors will be analyzed by the generalized estimating equations (GEE) approach. The cost of the three care models will also be compared. Findings of this study can contribute to current knowledge and practice for elderly patients with DM recovering from hip-fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or older (this criterion is based on our previous NHRI-funded study: Intervention program for elderly patients with hip fracture, 2001-2003),
2. Diagnosed with DM,
3. Admitted to CGMH from its emergency room due to hip fracture, and
4. Living in northern Taiwan (i.e.,greater Taipei area, Keelung, Taoyuan, or Shin-Ju Province).

Exclusion Criteria:

1. Clinical diagnosis of Cancer
2. Can't communicate with researchers

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | 2 years

SECONDARY OUTCOMES:
Activities of Daily life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing L Shyu, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taiwan, Taipei, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330